CLINICAL TRIAL: NCT04691050
Title: Clinical and Radiologic Evaluation of Root Canal Filling With OrthoMTA in Primary Molars Without Successors
Brief Title: Endodontic Management of Primary Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Sümeyra Akkoç, Assistant Proffessor, Tokat Gaziosmanpasa University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-KAEK-103
Record Dates: First submitted 2020-12-25; First posted 2020-12-31 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2020-12

CONDITIONS: Endodontically Treated Teeth
Keywords: Primary teeth; Root canal filling; Fractal analysis
MeSH Terms: conditions — Tooth, Nonvital | interventions — mineral trioxide aggregate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OrthoMta (BioMTA) (Other): OrthoMTA was applied in primary molars without successors
  Interventions: Procedure: OrthoMTA (BioMTA)

INTERVENTIONS:
Procedure: OrthoMTA (BioMTA) — Primary second molars without successors in which traditional root canal treatment with gutta-percha could not be performed was treated with OrthoMTA

SUMMARY:
The purpose of this study was to describe the clinical and radiological outcome of root canal treatment with OrthoMTA in primary second molars without successors in which traditional root canal treatment with gutta-percha could not be performed.

DETAILED DESCRIPTION:
The study included 13 primary mandibular second molars with infected pulp and congenitally missing second premolars in which traditional root canal treatment with gutta-percha was contraindicated. Pulpectomy was performed in each tooth and the canals were filled with OrthoMTA. The clinical and radiological outcomes of the treatment were evaluated at 3, 6, 9, and 12 months. Fractal analysis was used to detect changes in the trabecular bone after the treatment. Repeated measures analysis of variance test and two independent t-tests were used to evaluate the data.

ELIGIBILITY:
Inclusion Criteria:

* Selected to be preserved after an orthodontic consultation
* Absence of permanent tooth germ under second primary molars
* Sensitivity to percussion and palpation, complaints of spontaneous or persistent pain
* Presence of irreversible pulpitis or pulp necrosis, and abscess or fistula, presence of pathological mobility,
* Presence of internal and external pathological root resorption
* Furcal lesions
* Presence of infection exceeding 1/3 of the root
* Pathological loss of substantial bone support
* Loss of periodontal attachment
* Contraindication of traditional root canal treatment

Exclusion Criteria:

* Presence of any systemic disorder
* Presence of any syndrome
* A history or suspicion of allergies
* Age <7 years,
* Teeth selected to be extracted after an orthodontic consultation
* A score of 1(-) or 2(--) according to the Frankl Behavior Scale
* Parents who refused treatment, children who refused to receive the intended treatment once it was initiated

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2020-06-06 (Actual)

PRIMARY OUTCOMES:
Clinical success rate | 3 months after root canal treatment
  Clinical evaluation of root canal treatment was performed 3 months after treatment using the present clinical criteria. The treatment was decided a clinical success if the tooth fulfilled the following criteria:(1) continued function of the tooth without recurrence of infection; (2) no sensitivity on percussion and palpation; and (3) healthy soft tissues without fistula, abscess, and inflammation of the gums.
Radiographic success rate | 3 months after root canal treatment
  Radiographic evaluation of root canal treatment was performed 3 months after treatment using periapical radiograhps. The treatment was decided to be radiographically successful if it demonstrated the following criteria: (1) decreased radiolucency in the furcation or periradicular region, (2) absence of a new lesion formation.
Clinical success rate | 6 months after root canal treatment
  Clinical evaluation of root canal treatment was performed 6 months after treatment using the present clinical criteria. The treatment was decided a clinical success if the tooth fulfilled the following criteria:(1) continued function of the tooth without recurrence of infection; (2) no sensitivity on percussion and palpation; and (3) healthy soft tissues without fistula, abscess, and inflammation of the gums.
Radiographic success rate | 6 months after root canal treatment
  Radiographic evaluation of root canal treatment was performed 6 months after treatment using periapical radiograhps. The treatment was decided to be radiographically successful if it demonstrated the following criteria: (1) decreased radiolucency in the furcation or periradicular region, (2) absence of a new lesion formation.
Clinical success rate | 9 months after root canal treatment
  Clinical evaluation of root canal treatment was performed 9 months after treatment using the present clinical criteria. The treatment was decided a clinical success if the tooth fulfilled the following criteria:(1) continued function of the tooth without recurrence of infection; (2) no sensitivity on percussion and palpation; and (3) healthy soft tissues without fistula, abscess, and inflammation of the gums.
Radiographic success rate | 9 months after root canal treatment
  Radiographic evaluation of root canal treatment was performed 9 months after treatment using periapical radiograhps. The treatment was decided to be radiographically successful if it demonstrated the following criteria: (1) decreased radiolucency in the furcation or periradicular region, (2) absence of a new lesion formation.
Clinical success rate | 12 months after root canal treatment
  Clinical evaluation of root canal treatment was performed 12 months after treatment using the present clinical criteria. The treatment was decided a clinical success if the tooth fulfilled the following criteria:(1) continued function of the tooth without recurrence of infection; (2) no sensitivity on percussion and palpation; and (3) healthy soft tissues without fistula, abscess, and inflammation of the gums.
Radiographic success rate | 12 months after root canal treatment
  Radiographic evaluation of root canal treatment was performed 12 months after treatment using periapical radiograhps. The treatment was decided to be radiographically successful if it demonstrated the following criteria: (1) decreased radiolucency in the furcation or periradicular region, (2) absence of a new lesion formation.

SECONDARY OUTCOMES:
Change of fractal dimension | 12 months after root canal treatment
  The fractal dimension value of the furcation area between before treatment and 12 months after treatment were compared.

CONTACTS AND LOCATIONS:
Overall Officials: Sümeyra Akkoç, Asst Prof, Principal Investigator — Kutahya Health Sciences University
Locations (1):
- Tokat Gaziosmanpasa Univercity, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bezgin T, Ozgul BM, Arikan V, Sari S. Root canal filling in primary molars without successors: Mineral trioxide aggregate versus gutta-percha/AH-Plus. Aust Endod J. 2016 Aug;42(2):73-81. doi: 10.1111/aej.12132. Epub 2015 Nov 4. PMID 26534871
- [Background] O'Sullivan SM, Hartwell GR. Obturation of a retained primary mandibular second molar using mineral trioxide aggregate: a case report. J Endod. 2001 Nov;27(11):703-5. doi: 10.1097/00004770-200111000-00013. PMID 11716086
- [Background] Tunc ES, Bayrak S. Usage of white mineral trioxide aggregate in a non-vital primary molar with no permanent successor. Aust Dent J. 2010 Mar;55(1):92-5. doi: 10.1111/j.1834-7819.2009.01181.x. PMID 20415918
- [Background] Durovic E, Belus D. [Treatment of periadenitis mucosa necrotica recurrens with triamcinolon]. Stomatol Zpr. 1969;15(1):38-43. No abstract available. Czech. PMID 5282393